CLINICAL TRIAL: NCT01015365
Title: Cementless One-stage Revision in Fast-track Setting of the Chronic Infected Hip Arthroplasty
Brief Title: Cementless One-stage Revision of the Chronic Infected Hip Arthroplasty
Acronym: CORIHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CORIHA
Record Dates: First submitted 2009-11-06; First posted 2009-11-18 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Infection; Hip Joint Replacement
Keywords: Chronic infected hip arthroplasty; Fast-track; One-stage cementless revision
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Surgical revision (Other): Surgical cementless One-stage revision of the chronic infected hip arthroplasty
  Interventions: Procedure: Cementless one-stage surgical revision

INTERVENTIONS:
Procedure: Cementless one-stage surgical revision — A Cementless one-stage surgical revision is to be performed for all included in the cohort.

SUMMARY:
The investigators hypothesise that cementless one-stage exchange revision surgery can be performed in patients with chronically infected hip replacement with substantial benefits for the patients, in terms of fast rehabilitation, low re-revision rates and good long term results.

ELIGIBILITY:
Inclusion Criteria:

* Patient with clinical signs of infection for more than 4 weeks, arising from total hip arthroplasty (primary and revision), resurfacing hip arthroplasty or hemi-hip arthroplasty
* Informed oral and written consent given

Exclusion Criteria:

* Life expectancy under 2 years
* Cognitive dysfunction
* Pre-operative unwillingness to receive blood
* Intravenous drug abuse
* Alcoholism
* Immunocompromised patients
* Patients receiving immunosuppressive medication
* Ongoing systemic inflammatory disease
* Poorly regulated diabetes mellitus
* Renal failure (requiring dialysis)
* Acute systemic inflammatory response syndrome with proven infection (sepsis)
* Signs of coexisting active long-term local infection (i.e. endocarditis)
* Previous two-stage revision of hip arthroplasty due to ipsilateral chronic infection (regardless of symptom free interval) or contralateral chronic infection (within the last 2 years).
* < 6 weeks since last surgery of the affected hip
* If definition of infection is not fulfilled: infection defined as Culture positive: ≥ 3 positive intraoperative cultures (tissue biopsies a.m. Kamme-Lindberg) Culture negative: < 3 positive intraoperative cultures (tissue biopsies a.m. Kamme-Lindberg) + Chronic fistula with history of previous or existing secretion or Positive cultures in pre-operatively joint fluid aspiration with other clinical signs of infection or Visual pus or purulent fluid during exchange procedure with clinical signs of infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2009-11; Primary Completion 2016-10 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
re-infection | 2 years

SECONDARY OUTCOMES:
Revision for other cause than infection | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Soballe, Prof. D.Msc., Study Chair — Lundbeckfoundation center for fast-track hip and knee surgery; Jeppe Lange, M.D., Principal Investigator — Lundbeckfoundation center for fast-track hip and knee surgery
Locations (8):
- Denmark (8):
  - Orthopaedic Center, Alborg sygehus, Aarhus Universityhospital, Aalborg
  - Orthopaedic department, Aarhus Universityhospital, Aarhus
  - Gentofte Hospital, Hellerup
  - Orthopaedic department, Hvidovre Hospital, Hvidovre
  - Regionalhospital Silkeborg, Silkeborg
  - Sønderborg Hospital, Sønderborg
  - Vejle Hospital, Vejle
  - Regional Hospital Viborg, Viborg